CLINICAL TRIAL: NCT01282905
Title: Impact of the Mucosal Detoxification Mechanism of Hydrogen Sulphide on the Oxidation Pathway of Butyrate in Ulcerative Colitis
Brief Title: Hydrogen Sulfide Detoxification and Butyrate Metabolism in Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Prof. Kristin Verbeke, KULeuven
Other Study IDs: ML3999
Record Dates: First submitted 2011-01-24; First posted 2011-01-25 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — colon tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls
- Ulcerative colitis

SUMMARY:
The purpose of this study is to evaluate the relation between sulphide detoxification and butyrate metabolism at the level of gene expression and enzyme activity in ulcerative colitis patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

- Ulcerative colitis patients: patients diagnosed with ulcerative colitis

Exclusion Criteria:

* Healthy controls: no diagnosis of inflammatory bowel diseases
* Intake of antibiotics in the last month before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: IBD patients clinic (Universitaire Ziekenhuizen Leuven)
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2008-10; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, PhD, Principal Investigator — KU Leuven
Locations (1):
- KULeuven, Leuven, Belgium